CLINICAL TRIAL: NCT04701775
Title: A Randomized Double-Blind Controlled Trial of Lactobacillus Acidophilus Plus Bifidobacterium Animalis Subsp.Lactis, Versus Lactobacillus Rhamnosus GG Versus Placebo in Patients With Hypercholesterolemia
Brief Title: Effect of Different Probiotic Strains in Hypercholesterolemic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gözde Okburan, Assistant. Prof. Dr., Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/60-26
Record Dates: First submitted 2020-12-09; First posted 2021-01-08 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Hyperlipidemias
Keywords: serum lipids; hyperlipidemia; probiotics
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactobacillus rhamnosus GG Group (Experimental): Participants received only 1x106 cfu Lactobacillus rhamnosus GG once a day for 8 weeks.
  Interventions: Dietary Supplement: Only Lactobacillus rhamnosus GG strains
- Combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis Group (Experimental): Participants recevied a combined Lactobacillus acidophilus 1x109 cfu and Bifidobacterium animalis subsp.lactis 1x109 cfu once a day for 8 weeks.
  Interventions: Combination Product: Combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis strains
- Placebo (Placebo Comparator): Those participants received placebo capsule once a day for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Only Lactobacillus rhamnosus GG strains — 1x106 colony forming unit (CFU) Lactobacillus rhamnosus GG probiotic capsule
  Arms: Lactobacillus rhamnosus GG Group
Combination Product: Combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis strains — combination of Lactobacillus acidophilus 1x109 CFU and Bifidobacterium animalis subsp.lactis 1x109 CFU probiotic capsule
  Arms: Combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis Group
Other: Placebo — Placebo probiotic capsule
  Arms: Placebo

SUMMARY:
Regular probiotic use for 8 weeks was evaluated in individual with mild to moderate hyperlipidemia. Current study have been determined the use of different probiotics strains on lipid parameters such as; total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride levels as well as glycemic parameters such as; glucose, insulin, HOMA-IR levels. Also, hs-CRP levels were investigated as inflammatory parameter.

DETAILED DESCRIPTION:
In the light of recent studies, it has been shown that probiotics may have positive effects on hyperlipidemia. The aim of this study was to investigate the effect of probiotics mainly on blood lipids as well as homocysteine levels, glycemic control parameters and hs-CRP levels A randomized, double-blind placebo-controlled study was completed with a total of 51 individuals who have diagnosed with hyperlipidemia. Participants were randomly assigned into 3 groups according to the probiotic type they would consume, groups were as follows; Lactobacillus (probiotic group I) (n=18), Lactobacillus and Bifidobacterium (probiotic group II) (n=17) and placebo group (n= 16). They were all requested to have placebo or probiotic capsules every day for 8 weeks. Total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride levels were investigated as lipid metabolism parameters while fasting blood glucose, insulin, HOMA-IR levels were investigated as glycemic parameters. Also, hs-CRP levels were investigated as inflammatory parameter.

ELIGIBILITY:
Inclusion Criteria:

• Had a repeated total cholesterol level ≥200 mg/dL prior to allocate to the study group and to declined conventional lipid lowering medical treatment

Exclusion Criteria:

* Those with any chronic conditions other than hypercholesterolemia,
* Individuals with inherited lipid metabolic disorders,
* Individuals with chronic gastrointestinal disease,
* Individuals with immunodeficiency,
* Individuals with malignancy,
* Individuals with mental disabilities,
* Patients currently using any lipid lowering drugs, or an alternative treatment to lower blood cholesterol (such as probiotics) and individuals who have used antibiotics in the previous three months prior to study and
* Pregnant or lactating women were excluded from the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total cholesterol level with the use of combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis capsules at week 8 | Baseline and Week 8
  Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis decreases total cholesterol level. Change = (Baseline total cholesterol-Week 8 total cholesterol)
Change from baseline in Low Density Lipoprotein (LDL) levels with the use of combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis capsules at week 8 | Baseline and Week 8
  Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis decreases LDL cholesterol. Change = (Baseline LDL cholesterol values -Week 8 LDL cholesterol values)
Change from baseline in Triglyceride levels with the use of combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis capsules at week 8 | Baseline and Week 8
  Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis decreases triglyceride levels. Change = (Baseline triglyceride values -Week 8 triglyceride values)
Change from baseline in fasting glucose levels with the use of combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis capsules at week 8 | Baseline and Week 8
  Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis decreases fasting blood glucose levels. Change = (Baseline fasting glucose values -Week 8 fasting glucose values)
Change from baseline in fasting insulin levels with the use of combined Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis capsules at week 8 | Baseline and Week 8
  Lactobacillus acidophilus and Bifidobacterium animalis subsp.lactis decreases fasting insulin levels. Change = (Baseline fasting insulin values -Week 8 fasting insulin values)

SECONDARY OUTCOMES:
Change from baseline in total cholesterol level with the use of only Lactobacillus rhamnosus GG microorganism capsules at week 8 | Baseline and Week 8
  Lactobacillus rhamnosus GG microorganisms decreases total cholesterol level. Change = (Baseline total cholesterol-Week 8 total cholesterol)
Change from baseline in LDL cholesterol level with the use of only Lactobacillus rhamnosus GG microorganism capsules at week 8 | Baseline and Week 8
  Lactobacillus rhamnosus GG microorganisms decreases LDL cholesterol level. Change = (Baseline LDL cholesterol-Week 8 LDL cholesterol)
Change from baseline in triglyceride level with the use of only Lactobacillus rhamnosus GG microorganism capsules at week 8 | Baseline and Week 8
  Lactobacillus rhamnosus GG microorganisms decreases triglyceride level. Change = (Baseline triglyceride values-Week 8 trgylceride values)
Change from baseline in fasting glucose level with the use of only Lactobacillus rhamnosus GG microorganism capsules at week 8 | Baseline and Week 8
  Lactobacillus rhamnosus GG microorganisms decreases fasting glucosel level. Change = (Baseline fasting glucosel-Week 8 fasting glucose)
Change from baseline in fasting insulin with the use of only Lactobacillus rhamnosus GG microorganism capsules at week 8 | Baseline and Week 8
  Lactobacillus rhamnosus GG microorganisms decreases fasting insulin level. Change = (Baseline fasting insulin-Week 8 fasting insulin)

OTHER OUTCOMES:
Change from baseline in total cholesterol level with the use of placebo at week 8 | Baseline and Week 8
  Placebo capsules usually do not improve total cholesterol. Change = (Baseline total cholesterol values - Week 8 total cholesterol values)
Change from baseline in LDL cholesterol level with the use of placebo at week 8 | Baseline and Week 8
  Placebo capsules usually do not improve LDL cholesterol. Change = (Baseline LDL cholesterol values - Week 8 LDL cholesterol values)
Change from baseline in triglyceride level with the use of placebo at week 8 | Baseline and Week 8
  Placebo capsules usually do not improve triglyceride levels. Change = (Baseline triglyceride values - Week 8 total triglyceride values)
Change from baseline in fasting glucose level with the use of placebo at week 8 | Baseline and Week 8
  Placebo capsules usually do not improve fasting glucose levels. Change = (Baseline fasting glucose values - Week 8 total fasting glucose values)
Change from baseline in fasting insulin level with the use of placebo at week 8 | Baseline and Week 8
  Placebo capsules usually do not improve fasting insulin levels. Change = (Baseline fasting insulin values - Week 8 fasting insulin values)

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Okburan, Principal Investigator — Eastern Medittanean University
Locations (1):
- Gözde Okburan, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided